CLINICAL TRIAL: NCT01728428
Title: A Multicenter, Observational Study to Evaluate Clinical Manifestation, Diagnosis and Treatment of Primary Hemifacial Spasm in Chinese Patients
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116414
Record Dates: First submitted 2012-11-13; First posted 2012-11-19 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Hemifacial Spasm
Keywords: hemifacial spasm; observational study; clinical manifestation; treatment; Chinese
MeSH Terms: conditions — Hemifacial Spasm

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To determine the clinical manifestation, diagnosis and treatment options of primary hemifacial spasm in Chinese outpatient subjects

DETAILED DESCRIPTION:
About 1000 outpatient subjects will be recruited. The inclusion criteria include clinically diagnosed primary hemifacial spasm, male or female 18 to 80 years old and informed consent has been obtained. The exclusion criteria include secondary hemifacial spasm, other involuntary facial movement disorder, history of surgery of microvascular decompression of the facial nerve and so on. The outcome measures include the percentage of the treatment methods of HFS in outpatient subjects, aggrevated and relieved factors of HFS symptom, concomitant symptoms of HFS and adverse events of botulinum toxin treatment in HFS patients.

ELIGIBILITY:
Inclusion Criteria:

1.Clinically diagnosed primary hemifacial spasm

1. Tonic and clonic contractions of muscles innervated by the unilateral facial nerve.
2. No other neurological disorder. 2.Male or female 18 to 80 years old 3.Informed consent has been obtained

Exclusion Criteria:

1. Secondary hemifacial spasm: brainstem tumor, surgery, facial neuritis and so on.
2. Other involuntary facial movement disorder: facial synkinesia after facial palsy, tics, myokymia and focal motor seizures.
3. History of surgery of microvascular decompression of the facial nerve.
4. Participation in another clinical study currently.
5. Not able to understand and answer questionnaire.
6. Investigator's opinion that the subject has a concurrent condition(s) that may confound the study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 1000 Outpatient subjects from 15 centers across China.
Sampling Method: Probability Sample
Enrollment: 1003 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The percentage of the treatment methods of HFS in outpatient subjects | November, 2012

SECONDARY OUTCOMES:
Distribution of onset age of hemifacial spasm patients | November, 2012
Analysis of aggrevated and relieved factors of HFS symptom | November, 2012
Analysis of concomitant symptoms of hemifacial spasm | November, 2012
Adverse events of botulinum toxin treatment in hemifacial spasm | November, 2012

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Tan EK, Fook-Chong S, Lum SY, Lim E. Botulinum toxin improves quality of life in hemifacial spasm: validation of a questionnaire (HFS-30). J Neurol Sci. 2004 Apr 15;219(1-2):151-5. doi: 10.1016/j.jns.2004.01.010. PMID 15050451
- [Background] Wang A, Jankovic J. Hemifacial spasm: clinical findings and treatment. Muscle Nerve. 1998 Dec;21(12):1740-7. doi: 10.1002/(sici)1097-4598(199812)21:123.0.co;2-v. PMID 9843077
- [Background] Tan NC, Chan LL, Tan EK. Hemifacial spasm and involuntary facial movements. QJM. 2002 Aug;95(8):493-500. doi: 10.1093/qjmed/95.8.493. PMID 12145388
- [Background] Au WL, Tan LC, Tan AK. Hemifacial spasm in Singapore: clinical characteristics and patients ' perceptions. Ann Acad Med Singap. 2004 May;33(3):324-8. PMID 15175773
- [Result] Kenney C, Jankovic J. Botulinum toxin in the treatment of blepharospasm and hemifacial spasm. J Neural Transm (Vienna). 2008;115(4):585-91. doi: 10.1007/s00702-007-0768-7. Epub 2007 Jun 11. PMID 17558461